CLINICAL TRIAL: NCT06355297
Title: Educational Intervention Related to Pelvic Floor Care in Females in Sport
Brief Title: Educational Intervention Related to Pelvic Floor Care in Females in Sport: ACTITUD
Acronym: ACTITUD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Balearic Islands (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 124CER19.
Record Dates: First submitted 2024-03-31; First posted 2024-04-09 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-07

CONDITIONS: Pelvic Floor Disorders
Keywords: Female; Sport; Education
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Intervention Model Description: A quasiexperimental controlled trial is designed, with two arms: an experimental group and a control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Education about PF (Experimental): Education about PF. Participants will attend three 60-minutes educational online sessions.
  Interventions: Behavioral: Education about pelvic floor
- Control (No Intervention): Despite the fact that all females will be invited to participate in the study, those who did not attend the educational sessions will be considered as control group. These participants will not receive any educational session or information about PF prior to be evaluated.

INTERVENTIONS:
Behavioral: Education about pelvic floor — The three educational sessions will last 60 minutes, as follows: session1, anatomy of pelvic floor; session2, function and dysfunction of pelvic floor; session3, risk factor for pelvic floor dysfunctions.
  Arms: Education about PF

SUMMARY:
Pelvic floor dysfunctions (PFD) are especially prevalent among females who practice and compete in sport. One of the main reason is the great physical effort required to achieve the maximal sports performance. As conservational management, increasing the females' information is an important research line. However, gender stereotypes, embarrassment and normalization among females make it difficult to seek professional care. In this situation, prevention or management of PFD is limited.

New technologies could facilitate engaging virtual educational approaches. This study will evaluate the effects of an educational intervention compounded by three sessions (60 min of duration) with one week apart, about PFD, habits related with it, and existing gender stereotypes.

To this end, all female who practice and compete in any sport in Spain will be invited to attend an educational online intervention with theoretical-practical content about PFD. As eligibility criteria, participants should train and compete in any sport, and have federative license from regional or national sports federation at the moment of the start of the study. Participants should have at least 16 years old. The investigators expect 400 athletes to fulfill the questionnaires, of which the investigators expect 200 to attend the educational intervention. Before the educational intervention, all females will reply an anonymous questionnaire to inform about their knowledge of PFD, daily practices related to PFD, influencing gender stereotypes and PFD self-reported diagnosis. One month later, this questionnaire will be sent to females (both athletes who attended the educational intervention or not) to describe changes after attending the online educational intervention and compared to those females who did not attend it. The main outcomes will be the level of knowledge about PF, the number of habits potentially related to PFD, and score of gender stereotyped beliefs. As an additional outcome, it will be considered the PFD self-reported symptomatology.

DETAILED DESCRIPTION:
The educational intervention consisted on three 60-minutes online sessions, organized as follows:

Session 1: anatomical information about pelvic floor and exercises about pelvic floor consciousness; Session 2: function and dysfunction of pelvic floor and exercises related; Session 3: risk factor for pelvic floor dysfunctions and exercises to strengthen the pelvic floor musculature.

ELIGIBILITY:
Inclusion Criteria:

* To train and compete in any of the sport modality.
* To have federative license from a regional or national sport federation in the season when study starts.

Exclusion Criteria:

* Non applicable

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2024-04-09 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
Knowledge about pelvic floor | One month
  Change in the level of knowledge about pelvic floor according to the responses to an online questionnaire after attending the online educational sessions and compared to those females who do not attend educational sessions. To assess it, participants will reply an ad-hoc questionnaire with ten multiple-choice questions about pelvic floor structures. It will be counted the number of correct answers (0 points as the worst punctuation, 10 points as the best punctuation).
Habits related to pelvic floor dysfunctions | One month
  Change in number of habits that participants often carry out during their daily life, potentially related to pelvic floor dysfunctions, after attending the online educational sessions and compared to those athletes who do not attend educational sessions.

SECONDARY OUTCOMES:
Gender stereotypes beliefs | One month
  Change in the score related to gender stereotypes beliefs, after attending the online educational sessions and compared to those females who do not attend educational sessions. This score will be obtained after the sum of the factor1 and factor3 from the validated questionnaire CEGAFD (in English: beliefs and gender-based stereotypes concerning physical activity and sport). For the factor1 and factor3, females will rate from 1(completely disagree) to 4 (completely agree) to 7 and 5 gender stereotypes statements, respectively. The sum of the two factors will be the score of gender stereotypes beliefs (from 12 points as minimal gender stereotypes beliefs - 7 points for factor1 and 5 points for factor3 -, to 48 points as the maximal gender stereotypes beliefs - 28 points for factor1 and 20 points for factor3).
Occurrence of symptoms related to pelvic floor dysfunctions | One month
  It will be considered if pelvic floor dysfunction is self-reported through the questionnaire that athletes will reply. To this end, athletes will reply five yes-no questions regarding the occurrence of the main symptoms related to pelvic floor dysfunctions. In case of affirmative response in any of these diagnostic questions, it will be considered that this athlete has the symptom related to pelvic floor dysfunction. Between-group differences were considered.

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Romero-Franco, PhD, Principal Investigator — University of the Balearic Islands
Locations (1):
- University of the Balearic Islands, Palma de Mallorca, Balearic Islands, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goodridge SD, Chisholm LP, Heft J, Hartigan S, Kaufman M, Dmochowski RR, Stewart T, Reynolds WS. Association of Knowledge and Presence of Pelvic Floor Disorders and Participation in Pelvic Floor Exercises: A Cross-sectional Study. Female Pelvic Med Reconstr Surg. 2021 May 1;27(5):310-314. doi: 10.1097/SPV.0000000000000813. PMID 32217913
- [Background] Rashidi Fakari F, Hajian S, Darvish S, Alavi Majd H. Explaining factors affecting help-seeking behaviors in women with urinary incontinence: a qualitative study. BMC Health Serv Res. 2021 Jan 13;21(1):60. doi: 10.1186/s12913-020-06047-y. PMID 33435931
- [Background] Elenskaia K, Haidvogel K, Heidinger C, Doerfler D, Umek W, Hanzal E. The greatest taboo: urinary incontinence as a source of shame and embarrassment. Wien Klin Wochenschr. 2011 Oct;123(19-20):607-10. doi: 10.1007/s00508-011-0013-0. Epub 2011 Sep 22. PMID 21935649
- [Background] Reynolds WS, Kowalik C, Delpe SD, Kaufman M, Fowke JH, Dmochowski R. Toileting Behaviors and Bladder Symptoms in Women Who Limit Restroom Use at Work: A Cross-Sectional Study. J Urol. 2019 Nov;202(5):1008-1014. doi: 10.1097/JU.0000000000000315. Epub 2019 Oct 9. PMID 31059664